CLINICAL TRIAL: NCT02531841
Title: High-dose Chemotherapy and Autologous Stem Cell Transplant or Consolidating Conventional Chemotherapy in Primary CNS Lymphoma - Randomized Phase III Trial
Brief Title: High-dose Chemotherapy and ASCT or Consolidating Conventional Chemotherapy in Primary CNS Lymphoma
Acronym: MATRix
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Freiburg (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); International Extranodal Lymphoma Study Group (IELSG) (Other)
Responsible Party: Principal Investigator, Elisabeth Schorb, Medical Trial Coordinator, University Hospital Freiburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DRKS00005503
Record Dates: First submitted 2015-08-14; First posted 2015-08-25 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Diffuse Large B-cell-lymphoma
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Active Comparator): Induction Treatment 4 cycles MATRix (every 3 weeks), stem-cell harvest after 2nd cycle:
  * Rituximab 375 mg/m²/d i.v. (d0,5)
  * Methotrexate 3.5 g/m² i.v. (d1)
  * Cytarabine 2 x 2 g/m²/d i.v. (d2-3)
  * Thiotepa 30 mg/m² i.v. (d4)
  Consolidation Treatment 2 cycles of R-DeVIC (every 3 weeks):
  * Rituximab 375 mg/m²/d i.v. (d0)
  * Dexamethasone 40 mg/d i.v. (d1-3)
  * Etoposide 100 mg/m²/d i.v. (d1-3)
  * Ifosfamide 1500 mg/m²/d i.v. (d1-3)
  * Carboplatin 300 mg/m² i.v. (d1)
  Interventions: Drug: Arm A (Fortecortin®-ETOPOPHOS®-IFO-cell®-CARBO-cell®)
- Arm B (Active Comparator): Induction Treatment 4 cycles MATRix (every 3 weeks), stem-cell harvest after 2nd cycle:
  * Rituximab 375 mg/m²/d i.v. (d0,5)
  * Methotrexate 3.5 g/m² i.v. (d1)
  * Cytarabine 2 x 2 g/m²/d i.v. (d2-3)
  * Thiotepa 30 mg/m² i.v. (d4)
  Consolidation Treatment High-dose chemotherapy
  * Carmustine* 400 mg/m² i.v. (d-6)
  * Thiotepa 2 x 5 mg/kg/d i.v. (d-5-(-4))
  * Autologous Stem Cell Transplantation (d0)
    *if not available at study site, Busulfan can be administered instead:
  * Busulfan 3,2 mg/kg/d i.v. (d-8-(-7))
  * Thiotepa 2 x 5 mg/kg/d i.v. (d-5-(-4))
  * Autologous Stem Cell Transplantation (d0)
  Interventions: Drug: Arm B (TEPADINA®-CARMUBRIS®-Busilvex®)

INTERVENTIONS:
Drug: Arm A (Fortecortin®-ETOPOPHOS®-IFO-cell®-CARBO-cell®) — Arm A 4 cycles MATRix (every 3 weeks), stem-cell harvest after 2nd cycle:
  * Rituximab 375 mg/m²/d i.v. (d0,5)
  * Methotrexate 3.5 g/m² i.v. (d1)
  * Cytarabine 2 x 2 g/m²/d i.v. (d2-3)
  * Thiotepa 30 mg/m² i.v. (d4) Consolidation 2 cycles of R-DeVIC (every 3 weeks):
  * Rituximab 375 mg/m²/d i.v. (d0)
  * Dexamethasone 40 mg/d i.v. (d1-3)
  * Etoposide 100 mg/m²/d i.v. (d1-3)
  * Ifosfamide 1500 mg/m²/d i.v. (d1-3)
  * Carboplatin 300 mg/m² i.v. (d1)
  Other Names: Fortecortin®-ETOPOPHOS®-IFO-cell®-CARBO-cell®
  Arms: Arm A
Drug: Arm B (TEPADINA®-CARMUBRIS®-Busilvex®) — 4 cycles MATRix (every 3 weeks), stem-cell harvest after 2nd cycle:
  * Rituximab 375 mg/m²/d i.v. (d0,5)
  * Methotrexate 3.5 g/m² i.v. (d1)
  * Cytarabine 2 x 2 g/m²/d i.v. (d2-3)
  * Thiotepa 30 mg/m² i.v. (d4) Consolidation
  High-dose chemotherapy (HDT-ASCT):
  * Carmustine* 400 mg/m² i.v. (d-6)
  * Thiotepa 2 x 5 mg/kg/d i.v. (d-5-(-4))
  * Autologous Stem Cell Transplantation (d0)
    * if carmustine is not available at the investigation site, busulfan can be administered instead:
  * Busulfan 3,2 mg/kg/d (d-8-(-7))
  * Thiotepa 2 x 5 mg/kg/d i.v. (d-5-(-4))
  * Autologous Stem Cell Transplantation (d0)
  Other Names: TEPADINA®-CARMUBRIS®-Busilvex®
  Arms: Arm B

SUMMARY:
In the presently planned multicentre Phase III trial the two therapies will be compared: Patients will be randomized after intensified induction treatment with 4 cycles rituximab, methotrexate, cytarabine and thiotepa (MATRix) between first-line high-dose chemotherapy against conventional consolidating therapy with 2 cycles of conventional chemotherapy with R-DeVIC (rituximab, dexamethasone, etoposide, ifosfamide, carboplatin).

DETAILED DESCRIPTION:
Trial purpose and rationale Primary central nervous system lymphoma (PCNSL) is a highly aggressive disease with rising incidence over the past 30 years. Similar to other hematological diseases, the rationale for consolidation in PCNSL is the elimination of minimal residual disease. The efficacy of WBRT, which is the current standard for consolidation after HD-MTX-based systemic treatment, is being compared to HDT-ASCT in the ongoing IELSG-32 trial.

High-dose chemotherapy with carmustine or busulfan and thiotepa followed by autologous stem cell transplantation has been shown to be feasible and highly effective in newly diagnosed eligible patients, but also in the salvage situation.

The question we aim to answer is whether HDT-ASCT is superior to conventional therapy as consolidation after intensified immunochemotherapy in newly diagnosed PCNSL.

Rationale for this study:

Based on previously obtained good results from the treatment of recurrent or refractory PCNSL the DeVIC protocol was chosen for conventional consolidation treatment. This protocol, originally designed as a salvage protocol for aggressive NHL, crosses the blood-brain barrier and consists of multidrug resistant unrelated agents.

Treatment plan and procedure

Interventions

Induction treatment 4 cycles (every 3 weeks), stem-cell harvest after 2nd cycle:

* Rituximab 375 mg/m²/d i.v. (d 0,5)
* Methotrexate 3,5 g/m² i.v. (d1)
* Cytarabine 2 x 2 g/m²/d i.v. (d2-3)
* Thiotepa 30 mg/m² i.v. (d4)

Patients with PD after two cycles, SD/PD after four cycles of induction therapy or insufficient stem-cell harvest after three cycles are ineligible for randomization.

Consolidation Arm A 2 cycles of R-DeVIC (every 3 weeks):

* Rituximab 375 mg/m²/d i.v. (d0)
* Dexamethasone 40 mg/d i.v. (d1-3)
* Etoposide 100 mg/m²/d i.v. (d1-3)
* Ifosfamide 1500 mg/m²/d i.v. (d1-3)
* Carboplatin 300 mg/m² i.v. (d1)

Consolidation Arm B

High-dose chemotherapy (HDT-ASCT):

* Carmustine* 400 mg/m² i.v. (d-6)
* Thiotepa 2 x 5 mg/kg/d i.v. (d-5-(-4))
* Autologous Stem Cell Transplantation (d0)

  * if carmustine is not available at the investigation site, busulfan can be administered instead:
* Busulfan 3,2 mg/kg/d (d-8-(-7))
* Thiotepa 2 x 5 mg/kg/d i.v. (d-5-(-4))
* Autologous Stem Cell Transplantation (d0)

ELIGIBILITY:
Inclusion Criteria:

1. Immunocompetent patients with newly-diagnosed primary central nervous system B-cell lymphoma
2. Age 18-65 years irrespective of ECOG or 66-70 years (with ECOG Performance Status ≤2)
3. Histologically or cytologically assessed diagnosis of B-cell lymphoma by local pathologist.
4. Diagnostic sample obtained by stereotactic or surgical biopsy, CSF cytology examination or vitrectomy
5. Disease exclusively located in the CNS
6. At least one measurable lesion
7. Previously untreated patients (previous or ongoing steroid treatment admitted)
8. Sexually active patients of childbearing potential who agree to take adequate contraceptive measures during study participation
9. Written informed consent obtained according to international guidelines and local laws by patient or authorized legal representative in case patient is temporarily legally not competent due to his or her disease

ADDITIONAL RANDOMIZATION CRITERIA

1. Sufficient stem cell harvest (≥ 5 x 106 CD34+ cells/kg of body weight)
2. Complete remission, unconfirmed complete remission or partial remission
3. Central pathology results confirming local results

Exclusion Criteria:

1. Congenital or acquired immunodeficiency
2. Systemic lymphoma manifestation (outside the CNS)
3. Isolated ocular lymphoma without manifestation in the brain parenchyma or spinal cord
4. Previous or concurrent malignancies with the exception of surgically cured carcinoma in-situ of the cervix, carcinoma of the skin or other kinds of cancer without evidence of disease for at least 5 years
5. Previous Non-Hodgkin lymphoma at any time
6. Inadequate bone marrow (platelet count decreased ≥CTC grade 1, anemia ≥CTC grade 1, neutrophil count decreased ≥CTC grade 1), renal (creatinine clearance <60 ml/min), cardiac (ejection fraction decreased ≥CTC grade 2), or hepatic function (blood bilirubin increased ≥CTC grade 2, alanine aminotransferase increased ≥CTC grade 2, aspartate aminotransferase increased ≥CTC grade 2 or gamma-GT increased ≥CTC grade 2)
7. HBsAg, anti-HBc or HCV positivity
8. HIV infection, previous organ transplantation or other clinical evident form of immunodeficiency
9. Concurrent treatment with other experimental drugs or participation in a clinical trial within the last thirty days before the start of this study
10. Symptomatic coronary artery disease, cardiac arrhythmias uncontrolled with medication or myocardial infarction within the last 6 months (New York Heart Association Class III or IV heart disease)
11. Severe non-compensated pulmonary disease (IVC <55%, DLCO <40%)
12. Third space fluid accumulation >500 ml
13. Hypersensitivity to study treatment or any component of the formulation
14. Taking any medications likely to cause interactions with the study medication
15. Known or persistent abuse of medication, drugs or alcohol
16. Patient without legal capacity and who is unable to understand the nature, significance and consequences of the study and without designated legal representative
17. Persons who are in a relationship of dependency/employment to the sponsor and/ or investigator
18. Any familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
19. Concurrent (or planned) pregnancy or lactation
20. Fertile patients refusing to use safe contraceptive methods during the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2014-07; Primary Completion 2017-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure PFS will be measured by the number of events (PD, relapse or death from any cause) within the treatment arms | PFS is defined as the time from randomization until PD or relapse or death from any cause up to 24 months after end of treatment
  Progression-free survival PFS:
  Response Assessment III at the end of study treatment (EOT) visit and every imaging diagnostic assessments during follow-up period: during year 1-2: every 3 month

SECONDARY OUTCOMES:
The secondary outcome measure CR will be assessed on day 60 after randomization using the IPCG response criteria | CR will be determined on day 60 after randomization
  Response will be measured by the IPCG response criteria.
The secondary outcome measure Response duration will be measured by the time from CR, CRu or PR until relapse or PD using the IPCG response criteria | Time from CR, CRu or PR until relapse or PD up to 24 months after end of treatment
  Response duration observation times for patients where the event of interest was not observed, will be censored at the time last seen alive. Timepoints of evaluation are defined as every assessment during follow up period in accordance with the protocol.
  year 1-2: every 3 month
The secondary outcome OS is measured as time from randomization until death of any cause | OS is defined as time from randomization until death of any cause up to 24 months after end of treatment
  Timepoints of evaluation are defined as every assessment during follow up period in accordance with the protocol.
  year 1-2: every 3 month
Number of patients with (Serious) adverse events as assessed by CTCAE v4.0 | All SAEs that occur starting from the first administration of the study medication until day 60 after randomization.
  After this time period, only SAEs judged by the investigator to be related to at least one of investigational products will be reported
Number of patients with treatment related toxicity as assessed by CTCAE v4.0 | All toxicities that occur starting from the first administration of the study medication until day 60 after randomization.
  If an abnormal parameter is not listed in the toxicity table, an AE must be documented
Number of patients with neurotoxicity assessed by MMSE, EORTC QLQ-BN20 and the neuro-psychological battery | All parameters of neurotoxicity that occur starting from the first administration of the study medication up to 24 months after end of treatment.
  Timepoints of evaluation are defined as every assessment during follow up period in accordance with the protocol

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Illerhaus, PhD, Principal Investigator — Representative of Sponsor
Locations (2):
- Germany (2):
  - University Hospital Freiburg - Department for Hematology, Oncology and Stem cell Transplantion, Freiburg im Breisgau, Baden-Wurttemberg
  - Klinikum Stuttgart, Clinic of Hematology, Oncology and Palliative Care, Stuttgart Cancer Center / Tumor Center Eva Mayr-Stihl, Stuttgart, Baden-Wurttemberg

REFERENCES:
- [Result] Illerhaus G, Marks R, Ihorst G, Guttenberger R, Ostertag C, Derigs G, Frickhofen N, Feuerhake F, Volk B, Finke J. High-dose chemotherapy with autologous stem-cell transplantation and hyperfractionated radiotherapy as first-line treatment of primary CNS lymphoma. J Clin Oncol. 2006 Aug 20;24(24):3865-70. doi: 10.1200/JCO.2006.06.2117. Epub 2006 Jul 24. PMID 16864853
- [Result] Illerhaus G, Muller F, Feuerhake F, Schafer AO, Ostertag C, Finke J. High-dose chemotherapy and autologous stem-cell transplantation without consolidating radiotherapy as first-line treatment for primary lymphoma of the central nervous system. Haematologica. 2008 Jan;93(1):147-8. doi: 10.3324/haematol.11771. PMID 18166803
- [Result] Kasenda B, Schorb E, Fritsch K, Finke J, Illerhaus G. Prognosis after high-dose chemotherapy followed by autologous stem-cell transplantation as first-line treatment in primary CNS lymphoma--a long-term follow-up study. Ann Oncol. 2012 Oct;23(10):2670-2675. doi: 10.1093/annonc/mds059. Epub 2012 Apr 3. PMID 22473593
- [Result] Soussain C, Hoang-Xuan K, Taillandier L, Fourme E, Choquet S, Witz F, Casasnovas O, Dupriez B, Souleau B, Taksin AL, Gisselbrecht C, Jaccard A, Omuro A, Sanson M, Janvier M, Kolb B, Zini JM, Leblond V; Societe Francaise de Greffe de Moelle Osseuse-Therapie Cellulaire. Intensive chemotherapy followed by hematopoietic stem-cell rescue for refractory and recurrent primary CNS and intraocular lymphoma: Societe Francaise de Greffe de Moelle Osseuse-Therapie Cellulaire. J Clin Oncol. 2008 May 20;26(15):2512-8. doi: 10.1200/JCO.2007.13.5533. Epub 2008 Apr 14. PMID 18413641
- [Result] Motomura K, Natsume A, Fujii M, Ito M, Momota H, Wakabayashi T. Long-term survival in patients with newly diagnosed primary central nervous system lymphoma treated with dexamethasone, etoposide, ifosfamide and carboplatin chemotherapy and whole-brain radiation therapy. Leuk Lymphoma. 2011 Nov;52(11):2069-75. doi: 10.3109/10428194.2011.596967. Epub 2011 Jul 12. PMID 21745167
- [Derived] Schorb E, Finke J, Ferreri AJ, Ihorst G, Mikesch K, Kasenda B, Fritsch K, Fricker H, Burger E, Grishina O, Valk E, Zucca E, Illerhaus G. High-dose chemotherapy and autologous stem cell transplant compared with conventional chemotherapy for consolidation in newly diagnosed primary CNS lymphoma--a randomized phase III trial (MATRix). BMC Cancer. 2016 Apr 21;16:282. doi: 10.1186/s12885-016-2311-4. PMID 27098429